CLINICAL TRIAL: NCT02378246
Title: The Importance of Iodine During Pregnancy for Future Brain Function : a Randomized Placebo-controlled Trial. Swedish Iodine in Pregnancy and Development in Children (SWIDDICH) Study
Brief Title: Swedish Iodine in Pregnancy and Development in Children (SWIDDICH) Study
Acronym: SWIDDICH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13031305
Record Dates: First submitted 2015-01-19; First posted 2015-03-04 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Thyroid Gland; Node; Pregnancy; Cognitive Developmental Delay
Keywords: Iodine; Double-Blind Method; Randomized Controlled Tria; Cognitive Development
MeSH Terms: conditions — Thyroid Diseases | interventions — Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Tablet with vitamins and minerals, containing 150 ug iodine, 1 tablet daily (Experimental): Table of contents:
  Vitamin B2 1.4 mg, Vitamin B12 15 µg, Iron 12 mg, Zinc 12 mg, Iodine 150 µg, Selenium 50 µg, Calcium 250 mg
  Interventions: Dietary Supplement: Iodine
- Placebo: non-iodine containing multivitamin, 1 tablet daily (Placebo Comparator): Table of contents:
  Vitamin A 400 µg, Vitamin B1 1.4 mg, Vitamin B2 1.7 mg, Vitamin B6 1.8 mg, Vitamin B12 3 µg, Vitamin C 60 mg, Vitamin D 5 µg, Vitamin E 10 mg, Niacin 19 mg, Folic acid 200 µg
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iodine
  Arms: Tablet with vitamins and minerals, containing 150 ug iodine, 1 tablet daily
Dietary Supplement: Placebo
  Arms: Placebo: non-iodine containing multivitamin, 1 tablet daily

SUMMARY:
THE ULTIMATE GOAL of this project is to answer the question "In MILD IODINE DEFICIENCY (ID), should a tablet with vitamins and minerals, including 150 μg iodine/day be administered to pregnant women with a normal diet, to attain a normal cognitive development of the fetus or is there no cognitive deficit from mild ID and no extra iodine is needed?". To answer this question, the investigators planned a randomized, placebo-controlled trial of micronutrient supplementation during pregnancy in Sweden (SWIDDICH) with the follow-up of childrens' COGNITIVE DEVELOPMENT at 18 months, 3.5, 7 and 14 years.

Iodine deficiency (ID) is associated with thyroid morbidity and, especially in children, with impaired cognitive development. Sweden introduced iodine fortification of table salt 1936 and mental retardation due to severe ID is eradicated. Is mild ID during pregnancy also eradicated? If not, is this of importance? A national study performed by the investigators in 2007 showed iodine sufficiency in general population, but there are no pregnancy data. Local studies have raised concerns for mild ID during pregnancy in Sweden and a trans-sectional national study is currently ongoing.

The burning question for Sweden and the whole world is: is mild ID during pregnancy of importance for the developing brain of the fetus? Two large observational studies have shown association between mild ID during pregnancy and lower verbal IQ or educational performance at school-aged children. The world needs a randomized placebo-controlled trial (RTC) comparing the cognitive outcome in children exposed to mild ID during fetal life with children exposed to normal iodine levels during fetal life.

Our HYPOTHESIS is that pregnant women in Sweden have mild ID and that children exposed to mild ID during fetal life have a lower cognitive development, compared to children to mothers taking daily tablet with vitamins and minerals, including 150 ug iodine during pregnancy.

The MAIN AIM of the SWIDDICH trial is to determine if children exposed to deficient micronutrition including mild iodine deficiency (ID) during fetal life achieve worse cognitive development compared to children exposed to normal iodine status reached by maternal iodine supplementation.

DETAILED DESCRIPTION:
AIMS

* To determine if children exposed to deficient micronutrition including mild iodine deficiency (ID) during fetal life achieve worse cognitive development compared to children exposed to normal iodine status reached by maternal iodine supplementation.
* To investigate the interaction between iodine, selenium and iron, as components of the intervention.
* To compare urinary iodine concentration (UIC), thyroglobulin (Tg), free tetraiodothyronine (FT4) and thyroid stimulating hormone (TSH) in pregnant women on daily tablet with vitamins and minerals, including 150 µg iodine or placebo
* To compare milk iodine concentration (MIC) in colostrum, and TSH in the first 200 newborn children to pregnant women receiving daily tablet with vitamins and minerals, including 150 µg iodine or placebo

BACKGROUND Iodine deficiency increases the risk for hypothyroidism and goiter and during the pregnancy for abortion or cognitive and other abnormalities of the baby. According to the WHO recommendations, UIC during pregnancy should be 150-249 ug/L. In 2007 a national study showed iodine sufficiency in Swedish general population. It is debated whether or not iodine shall be given to pregnant women in iodine sufficient populations.

The research group started this randomized iodine intervention in pregnant women in 2012. The first hypothesis was that daily supplementation with a tablet with vitamins and minerals including 150 µg iodine is needed during pregnancy in Sweden in order to ensure normal iodine and thyroid hormone status in mothers and newborn children and that pregnant women in Sweden suffer from mild iodine deficiency (ID).

There is a substantial gap of knowledge with regards to whether mild ID during fetal life entails negative consequences on cognition. Two large observational studies have shown association between mild ID during pregnancy and lower IQ or educational performance in school-children. The only two randomized placebo-controlled trials (RCTs) studying mild ID in pregnancy were either too small for safe conclusions to be drawn ( Brucker-Davis et al, n=86), or did not manage to separate groups based on iodine levels (the MITCH study, Melse-Boonstra et al, n=839). The need for a RCT with sufficient sample size remains. This led the research team to form a second hypothesis within the trial: children exposed to deficient micronutrition including mild ID during fetal life have lower cognitive development compared to children to mothers taking a daily tablet with vitamins and minerals including150 ug iodine during pregnancy. The decision to expand the trial was made and the target number of participants to be recruited increased from 200 to 1275 in order to reach enough power to follow-up the childrens' cognitive development.

METHODS

Design

This is a prospective placebo-controlled trial of children whose mothers got iodine supplement 150 µg/day (a tablet with vitamins and minerals) or placebo (a multivitamin preparation without minerals) during pregnancy (week 10±2 until delivery). The target number participants during pregnancy is 1275 to enable sufficient power in the children follow-up (n=788). The main outcome is intelligence quotient (IQ) at 3.5 year of age. Cognitive development in children will be also assessed at 18 months, 7, and 14 years.

Pregnancy part

Pregnant women from more than ten maternity care centers in Sweden are randomized to daily receive a multivitamin tablet with minerals, including 150 µg iodine or placebo (multivitamin without iodine). The intervention starts at pregnancy week 8-12 and ends directly post-partum for the first 200 women and at pregnancy week 36±2weeks for the remaining participants. This time point may be adjusted to local circumstances, depending on when during the third trimester the routine visit at maternity care center takes place. Participants are included after the first visit by a midwife. Urine sample for UIC and U-creatinine, and blood sample for thyroid hormones, thyroid stimulating hormone (TSH), thyroglobuline (Tg) and thyroperoxidase antibodies (TPO-ab) are collected and a simple questionnaire is filled in at week 10±2 weeks of pregnancy and placebo/intervention is started. Selenium and iron are also measured. The same measurements are collected in week 25±1 week and week 36±2 weeks. Directly after delivery (within 5 days), MIC and UIC in the first 200 mother as well as UIC and TSH in their newborn child were collected and a simple questionnaire is filled in. Weight, length and APGAR in the child and pregnancy complications are registered. Blood is also frozen for future analyses and access to medical files is accepted.

In parallel 90 healthy female controls from Skaraborg area stratified for age and smoking habits are collected from a randomized sample attained by the Swedish Tax Agency. UIC, u-creatinine, FT4, TSH, Tg, TPO-ab, and samples to be frozen are collected and a questionnaire is filled in. Selenium and iron will be analyzed in blood sample from the first 200 pregnant women and from controls. The primary purpose for having a control population is to ascertain that the normal population in the area of Skaraborg is iodine sufficient.

Children follow-up

At 18 months ± 1 month psychomotor development is assessed by means of ASQ (Ages and Stages Questionnaire). At 3,5 years ± 2 months the IQ is measured (WPPSI-IV), behavior is assessed (CBCL questionnaire) and urine is collected for UIC measurement. At 7 years ± 3 months the following are assessed: IQ (WISC IV), motor development (Movement ABC), behavior (CBCL), symptoms related to attention deficit and hyperactivity disorder (ADHD, 5-15 Nordic questionnaire). Additionally, at 7 years ± 3 months urine is collected for UIC measurement, blood sample is taken for thyreoglobulin (Tg), thyroid hormones and deiodinases, and MRI of the brain is performed in a subsample. At 14 years ± 6 months all these, except for the Movement ABC, are repeated. On all occasions information on socio-economic status and other possible confounders are collected by means of questionnaires filled by parents and by children (14 years).

ELIGIBILITY:
PREGNANT WOMEN

Inclusion criteria

* Pregnant, week <13
* Age 18-40 years
* Intent of a full term pregnancy
* Agreement of taking no iodide containing supplements during the study except for study supplement

Exclusion Criteria

* Known current thyroid disease
* Risk factors for thyroid disease (history or heredity for thyroid, other autoimmune disease or symptoms of hypo-/hyperthyroidism) where the TSH is abnormal
* Possibility to not attend to the protocol according to the investigator's opinion
* Less than 6 months from previous pregnancy or lactating period
* Vegan

CONTROL WOMEN

Inclusion criteria

* Age 18-40 years
* Agreeing not to take iodide containing supplements 1 week prior to the collecting of the samples.

Exclusion criteria

* Current thyroid disease
* Risk factors for thyroid disease (history or heredity for thyroid or other autoimmune disease or symptoms of hypo-/hyperthyroidism) where the TSH is abnormal
* Possibility to not attend to the protocol according to the investigator's opinion
* Currently pregnant or lactating
* Less than 6 months from previous pregnancy or lactating period
* Vegans

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1337 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Intelligence quotient (IQ) at 3.5 years, WPPSI IV | when the child is at the age of 3,5 years ± 2 months
  Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition; IQ with sub-domains

SECONDARY OUTCOMES:
Psychomotor development at 18 months, ASQ-3 | when the child is at the age of 18 months ± 1 month
  Ages & Stages Questionnaire - Third Edition; a questionnaire filled in by parents
Intelligence quotient (IQ) at 7 years, WISC IV | when the child is at the age of 7 years ± 3 months
  Wechsler Intelligence Scale for Children - Fourth Edition; IQ with sub-domains
Intelligence quotient (IQ) at 14 years, WISC IV | when the child is at the age of 14 years ± 6 months
  Wechsler Intelligence Scale for Children - Fourth Edition; IQ with sub-domains
Behavioral problems at 3.5 years, CBCL | when the child is at the age of 3,5 years ± 2 months
  Child Behavior Checklist questionnaire filled in by parents
Behavioral problems at 7 years, CBCL | when the child is at the age of 7 years ± 3 months
  Child Behavior Checklist questionnaire filled in by parents
Behavioral problems at 14 years, CBCL | when the child is at the age of 14 years ± 6 months
  Child Behavior Checklist questionnaire filled in by parents
ADHD-related problems at 7 years, FTF | when the child is at the age of 7 years ± 3 months
  Nordic Questionnaire 5-15 (FTF) filled in by parents
ADHD-related problems at 14 years, FTF | when the child is at the age of 14 years ± 6 months
  Nordic Questionnaire 5-15 (FTF) filled in by parents
Motor skills at 7 years, Movement ABC | when the child is at the age of 7 years ± 3 months
  Movement ABC test performed by a physiotherapist
Brain development at 7 years, MRI | when the child is at the age of 7 years ± 3 months
  Magnetic Resonance Imaging; manual and automatic volumetry
Brain development at 7 years, MRI | when the child is at the age of 14 years ± 6 months
  Magnetic Resonance Imaging; manual and automatic volumetry
Urinary iodine concentration (UIC) in the mother, 1st trimester | 10±2 weeks (pregnancy)
Urinary iodine concentration (UIC) in the mother, 2nd trimester | 26±2 weeks (pregnancy)
Urinary iodine concentration (UIC) in the mother, 3rd trimester | 36±2 weeks (pregnancy)
Thyreoglobulin concentration in serum, in the mother, 1st trimester | 10±2 weeks (pregnancy)
Thyreoglobulin in serum, in the mother, 2nd trimester | 26±2 weeks (pregnancy)
Thyreoglobulin in serum, in the mother, 3rd trimester | 36±2 weeks (pregnancy)
Thyroid stimulating hormon concentration in serum, in the mother, 1st trimester | 10±2 weeks (pregnancy)
Thyroid stimulating hormon concentration in serum, in the mother, 2nd trimester | 26±2 weeks (pregnancy)
Thyroid stimulating hormon concentration in serum, in the mother, 3rd trimester | 36±2 weeks (pregnancy)
Free thyroxine concentration in serum, in the mother, 1st trimester | 10±2 weeks (pregnancy)
Free thyroxine concentration in serum, in the mother, 2nd trimester | 26±2 weeks (pregnancy)
Free thyroxine concentration in serum, in the mother, 3rd trimester | 36±2 weeks (pregnancy)
  Free thyroxine concentration, serum
Anti-TPO in the mother, 1st trimester | 10±2 weeks (pregnancy)
  Thyroid peroxidase antibody titer, plasma
Anti-TPO in the mother, 2nd trimester | 26±2 weeks (pregnancy)
  Thyroid peroxidase antibody titer, plasma
Anti-TPO in the mother, 3rd trimester | 36±2 weeks (pregnancy)
  Thyroid peroxidase antibody titer, plasma
B12 in the mother, 1st trimester | 10±2 weeks (pregnancy)
  Vitamin B12, serum
B12 in the mother, 2nd trimester | 26±2 weeks (pregnancy)
  Vitamin B12, serum
B12 in the mother, 3rd trimester | 36±2 weeks (pregnancy)
  Vitamin B12, serum
Selenium in the mother, 1st trimester | 10±2 weeks (pregnancy)
  Selenium, serum
Selenium in the mother, 2nd trimester | 26±2 weeks (pregnancy)
  Selenium, serum
Selenium in the mother, 3rd trimester | 36±2 weeks (pregnancy)
  Selenium, serum
Iron in the mother, 1st trimester | 10±2 weeks (pregnancy)
  Iron, serum
Iron in the mother, 2nd trimester | 26±2 weeks (pregnancy)
  Iron, serum
Iron in the mother, 3rd trimester | 36±2 weeks (pregnancy)
  Iron, serum
Milk iodine concentration (MIC) in colostrum | within 5 days after delivery
Urinary iodine concentration (UIC) in the newborn | within 5 days after delivery
Urinary iodine concentration (UIC) in the mother | within 5 days after delivery
Urinary iodine concentration (UIC) at 3.5 years | when the child is at the age of 3,5 years ± 2 months
Urinary iodine concentration (UIC) at 7 years | when the child is at the age of 7 years ± 3 months
Urinary iodine concentration (UIC) at 14 years | when the child is at the age of 14 years ± 6 months
Thyroid stimulating hormone, dry blood spot (DBS), in the newborn | within 5 days after delivery
TSH at 7 years | when the child is at the age of 7 years ± 3 months
  Thyroid stimulating hormone, dry blood spot (DBS)
TSH at 14 years | when the child is at the age of 14 years ± 6 months
  Thyroid stimulating hormone, dry blood spot (DBS)
TG at 7 years | when the child is at the age of 7 years ± 3 months
  Thyreoglobulin, dry blood spot (DBS)
TG at 14 years | when the child is at the age of 14 years ± 6 months
  Thyreoglobulin, dry blood spot (DBS)
FT4 at 7 years | when the child is at the age of 7 years ± 3 months
  Free thyroxine, dry blood spot (DBS)
FT4 at 14 years | when the child is at the age of 14 years ± 6 months
  Free thyroxine, dry blood spot (DBS)
Deiodinases at 7 years | when the child is at the age of 7 years ± 3 months
  Dry blood spot (DBS)
Deiodinases at 14 years | when the child is at the age of 14 years ± 6 months
  Dry blood spot (DBS)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson Nyström, Ass Prof, Principal Investigator — Center for Endocrinology and Metabolism, SAhlgrenska University Hospital
Locations (4):
- Sweden (4):
  - Umeå Universitet, Department of Clinical Sciences, Umeå, Västerbotten County
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skövde

IPD SHARING:
Plan to Share IPD: Undecided
This has not yet been discussed by the study group.

REFERENCES:
- [Derived] Manousou S, Eggertsen R, Hulthen L, Filipsson Nystrom H. A randomized, double-blind study of iodine supplementation during pregnancy in Sweden: pilot evaluation of maternal iodine status and thyroid function. Eur J Nutr. 2021 Sep;60(6):3411-3422. doi: 10.1007/s00394-021-02515-1. Epub 2021 Feb 23. PMID 33620551
- [Derived] Manousou S, Johansson B, Chmielewska A, Eriksson J, Gutefeldt K, Tornhage CJ, Eggertsen R, Malmgren H, Hulthen L, Domellof M, Nystrom Filipsson H. Role of iodine-containing multivitamins during pregnancy for children's brain function: protocol of an ongoing randomised controlled trial: the SWIDDICH study. BMJ Open. 2018 Apr 10;8(4):e019945. doi: 10.1136/bmjopen-2017-019945. PMID 29643159